CLINICAL TRIAL: NCT01642342
Title: A First-In-Human Phase I Study of sEphB4-HSA in Patients With Advanced Solid Tumors With Expansion at the Maximum Tolerated Dose (MTD) or Recommended Phase II Dose (RP2D).
Brief Title: Recombinant Albumin Fusion Protein sEphB4-HSA in Treating Patients With Metastatic or Recurrent Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Vasgene Therapeutics, Inc (Industry); The V Foundation for Cancer Research (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0C-11-3; NCI-2012-00971 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2012-07-14; First posted 2012-07-17 (Estimated); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Weekly Treatment (sEphB4-HSA) (Experimental): Patients receive recombinant albumin fusion protein sEphB4-HSA IV over 60 minutes on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: laboratory biomarker analysis; Other: pharmacological study; Biological: recombinant albumin fusion protein sEphB4-HSA
- Every 2 Weeks Treatment (sEphB4-HSA) (Experimental): Patients receive recombinant EphB4-HSA fusion protein IV over 60 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: laboratory biomarker analysis; Other: pharmacological study; Biological: recombinant albumin fusion protein sEphB4-HSA
- Every 3 Weeks Treatment (sEphB4-HSA) (Experimental): Patients receive recombinant EphB4-HSA fusion protein IV over 60 minutes on days 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: laboratory biomarker analysis; Other: pharmacological study; Biological: recombinant albumin fusion protein sEphB4-HSA

INTERVENTIONS:
Other: laboratory biomarker analysis — Correlative studies
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Biological: recombinant albumin fusion protein sEphB4-HSA — Given IV

SUMMARY:
This study is about an experimental drug called sEphB4-HSA (recombinant albumin fusion protein sEphB4-HSA). This research study will be the first time sEphB4-HSA is given to people. sEphB4-HSA prevents tumor cells from multiplying and blocks several compounds that promote the growth of blood vessels that bring nutrients to the tumor. sEphB4-HSA has shrunk colon, lung, breast, glioma, melanoma, prostate and Kaposi's sarcoma tumors in mice

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish the maximum tolerated dose (MTD) and recommended phase 2 dose (RP2D) of sEphB4-HSA.

II. To describe the dose limiting toxicities and adverse event profile of sEphB4-HSA in patients with advanced solid tumors.

III. To describe the pharmacokinetics of sEphB4-HSA. IV. To describe the anti-tumor activity of sEphB4-HSA as manifested by responses to treatment.

V. To obtain preliminary evaluation of effect of sEphB4-HSA on absolute circulating tumor cell (CTC) numbers as compared with pre-treatment levels using pre- and during treatment CTC. Exploratory evaluation of effect of sEphB4-HSA on downstream protein mediators of the Ephrin pathway (pAKT, pSrc) and their transcriptional target genes (rgs5 and psenen) will be performed.

VI. To collect pilot information to identify a dose or doses with biologic activity. Biologic activity after treatment with sEphB4-HSA will be defined as evidence of drug-on-target effect as manifested by reduction in absolute CTC numbers. Other exploratory evaluations of drug-on-target effect such as increase in transcript levels of psenen or rgs5 may be considered in the assessment of biologic activity.

OUTLINE: This is a dose-escalation study. Patients will be assigned to receive recombinant EphB4-HSA fusion protein intravenously (IV) over 60 minutes in one of the following treatment schedules:

1. Weekly treatment - administered on days 1, 8, 15, and 22. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
2. Every 2 weeks treatment - administered on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
3. Every 3 weeks treatment - administered on day 1. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* For expansion Cohort A: Advanced (metastatic or recurrent) pathologically proven solid tumor which has not responded to standard therapy or which has progressed following standard therapy for advanced disease and/or for which no standard therapy is known to be effective. Measurable disease required.
* For expansion Cohort B: Advanced pathologically proven mutant KRAS non-small cell lung cancer (group 1), pancreatic cancer (group 2; documentation of KRAS mutation not required), mutant KRAS colorectal cancer (group 3), head and neck squamous cell carcinoma (group 4) mesothelioma (group 5), hepatocellular cancer (group 6), and biliary carcinoma (group 7). Measurable disease required.
* Must agree, as part of the informed consent, to provide blood and tumor samples for molecular correlates, pharmacokinetics and pharmacodynamics. Patients in expansion cohort A must have tumor sites that are accessible for tumor biopsy and must agree to undergo a pre-treatment and post-treatment biopsy. Patients in cohort B group 3 & 4 must have tumor sites that are accessible for tumor biopsy and must agree to undergo a pre-treatment and post-treatment biopsy.
* Must have an Eastern Cooperative Oncology Group (ECOG) performance score of 0-1
* Life expectancy of at least 12 weeks
* Patients or their legal representatives must be able to comprehend and provide written informed consent
* White blood count (WBC) >= 3,000/μl
* Absolute neutrophil count (ANC) >= 1,500/μl
* Platelet count >= 100,000/μl (except in hepatocellular carcinoma patients with portal hypertension for whom a platelet count of >= 70,000/μl is allowed)
* Serum creatinine =< 1.5 X upper limit of normal (ULN) for reference lab
* Creatinine Clearance of >= 60 (as calculated by Cockcroft-Gault formula
* Serum bilirubin =< 1.5 mg/dL
* Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) levels =< 3X the ULN for the reference lab (=< 5X the ULN if there is evidence of hepatic involvement by malignant disease)
* Recovered to grade 1 from the effects (excluding alopecia) of any prior therapy for their malignancies
* Women of childbearing potential (WOCBP) and male patients with WOCBP partner must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the last dose of investigational product in such a manner that the risk of pregnancy is minimized
* WOCBP must have a negative serum test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours prior to the start of study drug
* Patients with hepatitis B infection must be on appropriate antiviral therapy
* For cohort B, group 1: Non-small cell lung cancer:

  * Must have advanced non-small cell lung cancer with mutant KRAS
  * Must have failed a minimum of one previous line of chemotherapy for advanced disease
* For cohort B, group 2: Pancreatic cancer:

  * Must have failed a minimum of one previous line of therapy for advanced disease
* For cohort B, group 3: Colorectal cancer:

  * Must have colorectal adenocarcinoma that harbor a KRAS mutation
  * Must have failed a minimum of one previous line of chemotherapy
* For cohort B, group 4: Head and neck squamous cell cancer:

  * Must have failed a platinum based chemotherapy regimen that was administered for advanced disease with a palliative intent; patients treated with concurrent platinum agent and radiation as definitive therapy are not eligible unless they subsequently received another line of systemic therapy.
* For cohort B, group 5: Mesothelioma:

  * Must have histologically or cytologically proven diagnosis of malignant mesothelioma; both pleural and peritoneal mesothelioma are allowed
  * Must have failed a minimum of one previous line of systemic therapy for advanced disease
* For cohort B, group 6: Hepatocellular carcinoma:

  * Patients with hepatocellular carcinoma do not need to have histologic confirmation of disease as long as they meet the radiologic criteria for diagnosis of HCC (evidence of arterial phase enhancement with corresponding venous or delayed phase wash out).
  * Must have advanced disease that is not amenable for resection or transplantation, and that is not treatable with liver directed modalities such as radiofrequency ablation or transarterial chemoembolization
  * Patients are not required to have failed Sorafenib
* For cohort B, group 7: Gallbladder cancer or cholangiocarcinoma:

  * Must have failed a minimum of one previous line of systemic therapy for advanced disease. If patient has had decompression of the biliary tree within the last 14 days, stability of the bilirubin level needs to be confirmed with two measurements that are within 5 to 7 days of each other.

Exclusion Criteria:

* Undergoing or have undergone in the past 28 days any other therapy for their cancer, including radiation and adjuvant therapy
* Major systemic infection requiring antibiotics 72 hours or less prior to first dose of study drug
* Untreated central nervous system (CNS) metastases; patients whose CNS metastases have been treated by surgery or radiotherapy, who are no longer on corticosteroids, and who are neurologically stable may be enrolled in the dose escalation portion of the trial
* Have New York Heart Association (NYHA) class 3 or 4, myocardial infarction, acute coronary syndrome, diabetes mellitus with ketoacidosis or chronic obstructive pulmonary disease (COPD) requiring hospitalization in the preceding 6 months; or any other intercurrent medical condition that contraindicates treatment with sEphB4HSA or places the patient at undue risk for treatment related complications
* Any other condition, including mental illness or substance abuse, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results
* Pregnant or lactating
* On any dose of warfarin or are on full dose anticoagulation with other agents, including low molecular weight heparin, antithrombin agents, antiplatelet agents and full dose aspirin within 7 days prior to first dose of study drug; patients on prophylactic doses of low-molecular weight heparin are allowed
* Any active bleeding in the last =< 4 weeks or have an otherwise known bleeding diathesis
* QTcF (Fridericia Correction Formula) > 480 on 2 out of 3 EKG's (if first EKG is < 480, no need to repeat, if first EKG is > 480 repeat twice for a total of 3 EKG's)
* For cohort B, group 1: Non-small cell lung cancer:

  * Must not have clinically significant active hemoptysis
* For cohort B, group 4: Head and neck squamous cell cancer:

  * Must not have evidence of major vessel involvement or encasement by tumor
* For cohort B, group 6: Hepatocellular Carcinoma:

  * Child Pugh score > 7
  * Ascites that is not medically controlled or that required a therapeutic paracentesis within last 3 months
  * Any episode of hepatic encephalopathy within the previous 6 months
  * Variceal bleeding within last 6 months
  * Patients with evidence of portal hypertension must have had an EGD within last year with appropriate treatment of esophageal varices as per standard of care

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2012-09-06 (Actual); Primary Completion 2019-05-29 (Actual); Study Completion 2019-05-29 (Actual)

PRIMARY OUTCOMES:
Toxicities observed at each dose level utilizing the National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version 4.0 | At least 4 weeks after the start of the first course
  Summarized in terms of type (organ affected or laboratory determination such as absolute neutrophil count), severity (by CTCAE and nadir or maximum values for the laboratory measures), time of onset (i.e. course number), duration, and reversibility or outcome. Tables will be created to summarize toxicities and side effects by dose and by course.
Number of patients with complete response (CR), partial response (PR), stable disease (SD), progressive disease (PD), or inevaluable (IE) | Up to 2 years
  Summarized by dose level in the dose escalation and in the expansion cohort.
Survival | Up to 2 years
  Summarized with Kaplan-Meier plots to describe the outcome.
Time to failure | Up to 2 years
  Summarized with Kaplan-Meier plots to describe the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony El-Khoueiry, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States